CLINICAL TRIAL: NCT05121935
Title: MAL-ED Metabolic: A Follow-Up of Chronic Disease at Puberty
Status: Not yet recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Haydom Lutheran Hospital (Other)
Responsible Party: Principal Investigator, Mark D. DeBoer, MD, MSc., MCR, Professor of Pediatrics, Division of Pediatric Endocrinology, University of Virginia
Other Study IDs: 200340
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Growth Failure; Intestinal Infection; Metabolic Syndrome; Glucose Intolerance
MeSH Terms: conditions — Failure to Thrive; Metabolic Syndrome; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect serum for later testing of markers of health, nutrition and inflammation, including C-reactive protein, IGF-1 and insulin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAL-ED cohort: Children initially followed from birth through 2 years old in the MAL-ED study (with some additional assessments in follow-up studies since then).

SUMMARY:
The concept that the roots of cardiometabolic disease start in early life was established by Dr. David Barker, who documented relationships between low birthweight (as a marker for challenges during gestation) and later cardiovascular disease (CVD). Later work has suggested that post-natal challenges (similar to prenatal ones) may also exhibit links to later cardiometabolic disease, with the strongest links appearing to be between low weight in early childhood and later hypertension and high waist circumference (WC). However, assessments for the relationship between early childhood challenges and insulin resistance and glucose regulation have been lacking and long-term cohort studies are few. In this project, we aim to assess children initially followed as part of The Etiology, Risk Factors, and Interactions of Enteric Infections and Malnutrition and the Consequences for Child Health (MAL-ED) study, where they received frequent measures of anthropometry and laboratory assessments for intestinal pathogens. These children are now of peri-pubertal age--a time period associated with metabolic shifts. We will assess for glucose dysregulation and findings associated with the metabolic syndrome, and we will analyze potential associations between current chronic disease risk findings with early life poor growth and intestinal pathogen carriage rate. As such, we hope to uncover potential targets in early life health to reduce later chronic disease risk.

DETAILED DESCRIPTION:
The relationship between prenatal challenges and later risk for chronic disease has been well established. Our group previously assessed the hypothesis that post-natal challenges (similar to prenatal ones) would exhibit links to later cardiometabolic disease. This was performed using retrospective data from a long-term cohort of children in Guatemala, demonstrating novel findings that higher degrees of diarrhea burden in the first 6 months of life (as a marker of nutritional and/or inflammatory stressors) were associated with a greater risk of metabolic syndrome as adults The causes of these findings are not known, though postulated mechanisms include epigenetic reprograming of metabolic rate, hormonal regulation and vascular tone. Unfortunately, long-term cohort studies are few, limiting opportunities to evaluate these links prospectively.

The Haydom Global Health Research Center in north central Tanzania represents an important rural setting for performing high-quality medical research in sub-Saharan Africa (5). The region around Haydom has a high degree of stunting and enteric pathogen carriage among a cohort of children followed in the area from 2009-2013 as part of the multi-country study "The Etiology, Risk Factors, and Interactions of Enteric Infections and Malnutrition and the Consequences for Child Health (MAL-ED)."

These children followed in Haydom during MAL-ED had monthly anthropometry and stool pathogen analysis, as well as extensive demographic data. This provides an opportunity to follow up on these children to assess for potential links between early life challenges (both enteric disease, infections and nutritional deficiencies) and later chronic disease risk, including lipid abnormalities, glucose intolerance and blood pressure elevations. The current proposal is to follow up on these children at the age of typical entry into puberty, as this is a common shift in metabolism when many children begin to exhibit metabolic abnormalities. We will assess these children for multiple measures:

* Anthropometry (height, weight, BMI, waist circumference)
* Assessment of pubertal stage by exam or questionnaire
* Blood pressure
* Lipids (LDL, HDL, triglycerides)
* CRP
* Oral glucose tolerance test (OGTT)
* Fasting insulin
* Metabolic syndrome (MetS) severity score
* Blood saved for future epigenetic testing

We will use linear and and logistic regression to determine associations between 1) mean number of monthly pathogens (individual pathogens and in aggregate) and 2) reported symptoms (fever, cough, diarrhea), with multiple MetS-related outcomes: BMI percentile, WC, fasting insulin, 2-hour glucose following OGTT, triglycerides, HDL cholesterol, normalized BP and a MetS diagnosis.

The underlying hypothesis is that there will be consistent links between features of MetS (in particular blood pressure, waist circumference and insulin resistance) with 1) enteric pathogen burden (overall and for particularly virulent pathogens such as Enterotoxigenic E.coli) and 2) poor early life growth.

ELIGIBILITY:
Inclusion Criteria:

* Participated in original MAL-ED cohort

Exclusion Criteria:

* Did not participate in original MAL-ED cohort

Ages: 9 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: This is a follow-up study of children who were originally in the MAL-ED cohort.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Current Systolic BP--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current systolic BP z-score vs. number enteric pathogens by age 2 years (from MAL-ED)

SECONDARY OUTCOMES:
Current Systolic BP--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current systolic BP z-score vs. BMI z-score at age 2 years (from MAL-ED), adjusted for current BMI z-score
Current Diastolic BP--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current diastolic BP z-score vs. number enteric pathogens by age 2 years (from MAL-ED)
Current Diastolic BP--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current diastolic BP z-score vs. BMI z-score at age 2 years (from MAL-ED), adjusted for current BMI z-score
Current BMI z-score--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current BMI z-score vs. number enteric pathogens by age 2 years (from MAL-ED)
Current waist circumference--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current waist circumference vs. number enteric pathogens by age 2 years (from MAL-ED)
Metabolic syndrome (MetS) severity score--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current MetS severity z-score vs. number enteric pathogens by age 2 years (from MAL-ED)
Current metabolic syndrome (MetS) severity score--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current MetS severity z-score vs. number enteric pathogens by age 2 years (from MAL-ED), adjusted by current waist circumference
Current glucose from oral glucose tolerance test (OGTT) at 2 hours--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current 2-hour OGTT glucose vs. number enteric pathogens by age 2 years (from MAL-ED)
Current glucose from oral glucose tolerance test (OGTT) at 2 hours--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current 2-hour OGTT glucose vs. BMI z-score at age 2 years (from MAL-ED), adjusted by current BMI z-score
Current fasting triglycerides--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current ln(triglycerides) vs. number enteric pathogens by age 2 years (from MAL-ED)
Current fasting triglycerides--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current ln(triglycerides) vs. BMI z-score at age 2 years (from MAL-ED), adjusted by current BMI z-score
Current HDL cholesterol--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current HDL cholesterol vs. number enteric pathogens by age 2 years (from MAL-ED)
Current HDL cholesterol--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current HDL cholesterol vs. BMI z-score at age 2 years (from MAL-ED), adjusted by current BMI z-score
Current fasting glucose--relationship to number of enteric pathogens by age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current fasting glucose vs. number enteric pathogens by age 2 years (from MAL-ED)
Current fasting glucose--relationship to BMI z-score at age 2 years | Measured during current study (1 year +/- 3 months)
  Regression analysis of current fasting glucose vs. BMI z-score at age 2 years (from MAL-ED), adjusted by current BMI z-score

CONTACTS AND LOCATIONS:
Overall Officials: Mark D DeBoer, MD, Principal Investigator — University of Virginia; Estomih Mduma, MPH, Study Director — Haydom Global Health Research Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeBoer MD, Lima AA, Oria RB, Scharf RJ, Moore SR, Luna MA, Guerrant RL. Early childhood growth failure and the developmental origins of adult disease: do enteric infections and malnutrition increase risk for the metabolic syndrome? Nutr Rev. 2012 Nov;70(11):642-53. doi: 10.1111/j.1753-4887.2012.00543.x. PMID 23110643
- [Background] DeBoer MD, Chen D, Burt DR, Ramirez-Zea M, Guerrant RL, Stein AD, Martorell R, Luna MA. Early childhood diarrhea and cardiometabolic risk factors in adulthood: the Institute of Nutrition of Central America and Panama Nutritional Supplementation Longitudinal Study. Ann Epidemiol. 2013 Jun;23(6):314-20. doi: 10.1016/j.annepidem.2013.03.012. Epub 2013 Apr 19. PMID 23608305
- [Background] Mduma ER, Gratz J, Patil C, Matson K, Dakay M, Liu S, Pascal J, McQuillin L, Mighay E, Hinken E, Ernst A, Amour C, Mvungi R, Bayyo E, Zakaria Y, Kivuyo S, Houpt ER, Svensen E. The etiology, risk factors, and interactions of enteric infections and malnutrition and the consequences for child health and development study (MAL-ED): description of the Tanzanian site. Clin Infect Dis. 2014 Nov 1;59 Suppl 4:S325-30. doi: 10.1093/cid/ciu439. PMID 25305305
- [Background] Scharf RJ, Rogawski ET, Murray-Kolb LE, Maphula A, Svensen E, Tofail F, Rasheed M, Abreu C, Vasquez AO, Shrestha R, Pendergast L, Mduma E, Koshy B, Conaway MR, Platts-Mills JA, Guerrant RL, DeBoer MD. Early childhood growth and cognitive outcomes: Findings from the MAL-ED study. Matern Child Nutr. 2018 Jul;14(3):e12584. doi: 10.1111/mcn.12584. Epub 2018 Feb 2. PMID 29392824
- [Derived] Nemati K, Michael YZ, Hhando BP, Jatosh S, Houpt ER, Mduma E, DeBoer MD. Catch-up growth following early-life stunting in a low-resource area in rural Tanzania: the MAL-ED Metabolic study. BMJ Open. 2025 Aug 21;15(8):e100955. doi: 10.1136/bmjopen-2025-100955. PMID 40840991